CLINICAL TRIAL: NCT06573749
Title: Effect of 12-week Bioactive Whey Protein Concentrate Supplementation on the Neuromuscular System of Healthy, Recreationally Active Adults
Brief Title: Effect of 12-week Milk Fat Globule Membrane Supplementation on the Human Muscle Function of Healthy, Recreationally Active Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loughborough University (Other)
Collaborators: Volac International Limited (Unknown)
Responsible Party: Principal Investigator, Edward Sadula, Doctoral Researcher, Loughborough University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 16406
Record Dates: First submitted 2024-08-21; First posted 2024-08-27 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Ageing Well; Neuromuscular Function
Keywords: Nutrition; Neuromuscular; Milk fat globule membrane

STUDY DESIGN:
Intervention Model Description: Participants will be allocated to one of two groups, placebo or bioactive whey protein concentrate supplement. Within each supplement group there will be 2 age subgroups (young and older).
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The placebo and bioactive whey protein concentrate supplement have been given specific codes by an external investigator to ensure that the participant and investigator are blinded. The external investigator will reveal which code corresponds to which supplement group once the principal investigator has completed statistical analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bioactive whey protein concentrate supplement group (Experimental): This group will consume a supplement called bioactive whey protein concentrate, a whey protein concentrate that contains milk fat globule membrane.
  Interventions: Dietary Supplement: Bioactive whey protein concentrate
- Placebo group (Placebo Comparator): This group will consume an isocaloric, isonitrogenous whey protein isolate supplement that does not contain phospholipids or sphingomyelin. Dextrose has been added to the whey protein isolate to ensure the 2 supplements are isocaloric.
  Interventions: Dietary Supplement: Whey protein isolate supplement

INTERVENTIONS:
Dietary Supplement: Bioactive whey protein concentrate — Every day for 12 weeks, participants will mix 1 scoop of supplement with ~350ml of water and consume the resultant drink alongside their breakfast.
  Arms: Bioactive whey protein concentrate supplement group
Dietary Supplement: Whey protein isolate supplement — Every day for 12 weeks, participants will mix 1 scoop of supplement with ~350ml of water and consume the resultant drink alongside their breakfast.
  Arms: Placebo group

SUMMARY:
The main aim of this study is to understand if chronic supplementation (12 weeks) of a milk fat globule membrane containing supplement, called bioactive whey protein concentrate, improves human muscle function greater than a placebo supplement within a cohort of healthy, recreationally active adults. Furthermore, we aim to investigate whether any potential benefits of milk fat globule membrane are influenced by age through the assessment of 2 distinct age subgroups (young and older). We hypothesise that neuromuscular function (strength and power) will increase from pre to post within the group that consumes bioactive whey protein concentrate but not the placebo group, with a greater increase in the older group compared to the young group.

DETAILED DESCRIPTION:
Nutritional strategies, including supplementation, are widely sought after to improve the function of the neuromuscular system (muscle strength and power). Milk fat globule membrane (MFGM, composed of the membrane that surrounds milk fat droplets) has begun to receive increasing attention as a potential supplement to improve muscle function and size due to a series of promising longitudinal studies (> 4 weeks of supplementation), however the overall findings are still conflicting which is likely due to methodological limitations of previous studies. Therefore, it is important to thoroughly investigate whether chronic supplementation of a MFGM-containing supplement is effective at improving the function and physiology of the neuromuscular system within healthy, recreationally active adults.

This study aims to compare the effects of chronic (12 weeks) bioactive whey protein concentrate (BWPC) supplementation versus an isocaloric, isonitrogenous whey protein isolate placebo on the physiology (contractile properties, coactivation, timing of action potentials), morphology (total/functional muscle cross-sectional area/volume), and function of the neuromuscular system of healthy, recreationally active adults.

Utilising a randomised, double-blind, parallel group study design, participants will be allocated to one of two groups: BWPC or placebo supplement group. Once consented, participants will complete screening questionnaires to confirm their eligibility. Altogether, participants will be required to attend 5 laboratory sessions (1 familiarisation ~ 1.5 hours, 4 main measurement sessions each ~ 2 hours) at the neuromuscular laboratories situated within the Matthew Arnold building at Loughborough University. The familiarisation and first two baseline measurement sessions will be done over a 2-week period, after which participants will be asked to consume a supplement daily for 12 weeks (84 daily doses) while they maintain their usual lifestyle (diet and exercise/physical activity). Then they will attend two further post measurement sessions, with the first being at exactly 12 weeks of supplementation (i.e. 84th day) and the second being 3-4 days later (i.e. 87th or 88th day). The supplementation protocol will involve participants mixing 1 scoop of supplement with water and consuming the resultant drink alongside their breakfast. Participants will be required to fill in a diet record form twice across the supplementation period (week 3 and 9), which involves weighing and recording what they eat/drink over 3 consecutive days. Physical activity at pre and post will be assessed through the International Physical Activity Questionnaire (IPAQ, short format).

During the familiarisation session participants will get to try all of the types of contractions (voluntary and involuntary) to be performed in the main measurement sessions, but without the recording of electromyography (EMG). The first measurement session at baseline/post will begin with countermovement jumps on a force plate. The remainder of the session will involve various isometric knee extension or flexion contractions within a custom-built isometric dynamometer. This will include maximal and explosive voluntary contractions to assess maximal strength of the knee extensors and flexors and rate of force development of the knee extensors, respectively. Supramaximal femoral nerve stimulation will be utilised to evoke twitch contractions of the knee extensors. Submaximal transcutaneous muscle stimulation will be performed to assess the force-frequency relationship (1 - 100 Hz) of the knee extensors. Finally, submaximal knee extension contractions (10 and 25% of maximal voluntary force) will be performed while a concentric needle electrode is inserted into the vastus lateralis to assess the stability of neuromuscular junction transmission. Throughout this measurement session, surface EMG signals will be collected by placing surface EMG electrodes on each of the 3 superficial quadriceps muscles (rectus femoris, vastus lateralis and medialis) and on the hamstrings (medial and lateral).

Within the second measurement session at pre/post, participant's will have an 3.0 T MRI scan of the lower limbs. The procedure will be clearly explained to the participant before they sign the MRI agreement form and fill in the MRI safety questionnaire.

For this study we want to assess whether any potential benefits of milk fat globule membrane are influenced by age. Therefore, we will be recruiting 2 subgroups (young 18 - 30 years old; older 60 - 75 years old). The power analysis was based on detecting a group by time interaction for isometric strength, with input parameters of: effect size = 0.15, alpha = 0.05, power = 0.8, correlation among repeated measures = 0.8. Altogether, 38 participants are needed as a minimum within each age group (19 per group). However, to account for a 25% drop-out rate, 48 participants will be recruited for each age group. The total number of participants recruited will be 96 (48 young, 48 older).

Statistical analysis will involve fitting linear mixed effect models to detect any main effects or interactions, with supplement group, time (pre vs post), and their interaction as fixed effects, and participant as a random intercept. Visual plots (histograms and quantile-quantile plots) will be used to verify the assumptions of normality, linearity, and homoscedasticity of residuals.

ELIGIBILITY:
Inclusion Criteria:

* 18-30 or 60-75 years old
* Male or female
* Healthy with no contraindications to exercise
* Classified as recreationally active (meet the government's guidelines for weekly physical activity - 150 minutes of moderate physical activity or 75 minutes of vigorous physical activity)

Exclusion Criteria:

* Any injury, medical condition or symptom precluding the ability to complete strenuous exercise as identified by the health screen questionnaire and physical activity readiness questionnaire
* Uncontrolled hypertension (blood pressure of 140/90 mmHg or higher) as identified by recording resting blood pressure
* Neuromuscular or musculoskeletal disease
* Occurrence of a severe injury to the lower limbs or back within the previous 6 months (time loss of > 21 days of normal activity)
* Occurrence of a minor injury to the lower limbs or back within the previous month (time loss of >1 day of normal activity)
* Do not meet the government guidelines of minimum weekly physical activity as revealed by the IPAQ-SF
* Allergic to dairy or pea, or lactose intolerant
* Complete greater than 6 hours structured exercise per week as revealed by the exercise and physical activity form
* Consumption of supplements that may confound the results of the present study within the previous 3 months (includes any form of protein supplement, creatine, pre-workout supplements, any form of testosterone supplement, amino acids, beta-alanine, beta- hydroxy-beta-methylbutyrate (HMB), fish or krill oil, collagen supplements, any choline- containing supplement, or any phospholipid-containing supplement) as highlighted by the health screen questionnaire
* Taking anticoagulants or antiplatelet drugs
* Use of antidepressant/anti-anxiety medication
* Having a blood borne virus, or a partner who has a blood-borne virus
* Extreme diet classified as identified by the food-frequency questionnaire

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-03-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Maximal voluntary isometric torque of the knee extensors | 12 weeks
  Assessed during maximal voluntary contractions (Nm)

SECONDARY OUTCOMES:
Rate of torque development of the knee extensors | 12 weeks
  Assessed during explosive isometric contractions (Nm/s)
Peak twitch torque (knee extensors) | 12 weeks
  (Nm)
Time to peak twitch torque (knee extensors) | 12 weeks
  (ms)
Half-relaxation time during twitch contractions (knee extensors) | 12 weeks
  (ms)
Neural activation of the agonist (quadriceps) and antagonist (hamstrings) | 12 weeks
  Surface electromyography (root mean square amplitude)
Force-frequency relationship of the knee extensors | 12 weeks
  Peak torque across the various stimulation frequencies (1 - 100 Hz, Nm)
Neuromuscular junction transmission stability | 12 weeks
  Extraction of variables (e.g. jitter and jiggle) from the decomposition of intramuscular electromyography signals recorded during submaximal (10 and 25% of maximal voluntary force) isometric knee extension contractions held for 20 seconds
Cross-sectional area of upper leg muscles | 12 weeks
  Measured by MRI (cm^2)
Volume of upper leg muscles | 12 weeks
  Measured by MRI (cm^3)
Functional cross-sectional area of upper leg muscles | 12 weeks
  Measured by MRI (cm^2)
Functional volume of upper leg muscles | 12 weeks
  Measured by MRI (cm^3)
Intramuscular fat infiltration of upper leg muscles | 12 weeks
  Measured by MRI (% of intramuscular fat)
Neuromuscular power | 12 weeks
  Measured during countermovement jumps on a force plate (W)
Level of physical activity | 12 weeks
  International Physical Activity Questionnaire (IPAQ)
Habitual energy intake | 12 weeks
  Measured by food diary (kcal.day-1)
Habitual protein intake | 12 weeks
  Measured by food diary (g.day-1)
Habitual carbohydrate intake | 12 weeks
  Measured by food diary (g.day-1)
Habitual fibre intake | 12 weeks
  Measured by food diary (g.day-1)
Habitual fat intake | 12 weeks
  Measured by food diary (g.day-1)
Habitual choline intake | 12 weeks
  Measured by food diary (mg.day-1)
Maximum voluntary isometric torque of the knee flexors | 12 weeks
  Assessed during maximal voluntary contractions (Nm)

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sadula, BSc, MSc, Principal Investigator — Loughborough University
Locations (1):
- Loughborough University, Loughborough, Leicestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No